CLINICAL TRIAL: NCT02764021
Title: Cut Down on Carbohydrate Usage in the Diet of Type 2 Diabetes; Mechanisms of Effective Therapy of Diabetes by Selective Choice of Macronutrients. The Isoenergetic Study.
Brief Title: Cut Down on Carbohydrate Usage in the Diet of Type 2 Diabetes
Acronym: CutDM-iso
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University of Copenhagen (Other); University of Aarhus (Other)
Responsible Party: Principal Investigator, Mads Gustav Juul Skytte, MD, PhD student, Bispebjerg Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-15020386
Record Dates: First submitted 2016-04-26; First posted 2016-05-06 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: HbA1c; Diabetes-Releated Complications; Diet, Low Carbohydrate; Carbohydrate-Restricted Diet; Diabetes Mellitus; Metabolic Disorder; Glucose Metabolism Disorders; Endocrine System Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Metabolic Diseases; Glucose Metabolism Disorders; Endocrine System Diseases | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. (Experimental): Subjects will be randomly assigned to initially receive 6 weeks of standard antidiabetic dietary treatment or 6 weeks of experimental carbohydrate-restricted dietary treatment, crossing over to the opposite diet from week 6 to 12.
  Interventions: Dietary Supplement: Carbohydrate-Restricted Diet
- 2. (Active Comparator): Subjects will be randomly assigned to initially receive 6 weeks of standard antidiabetic dietary treatment or 6 weeks of experimental carbohydrate-restricted dietary treatment, crossing over to the opposite diet from week 6 to 12.
  Interventions: Dietary Supplement: Standard Antidiabetic Diet

INTERVENTIONS:
Dietary Supplement: Carbohydrate-Restricted Diet — Macronutritional composition: Carbohydrate 30 E%, Protein 30 E%, Fat 40 E%
  Arms: 1.
Dietary Supplement: Standard Antidiabetic Diet — Macronutritional composition: Carbohydrate 50 E%, Protein 13 E%, Fat 17 E%
  Arms: 2.

SUMMARY:
Scientific evidence for the dietary treatment of type 2 diabetes (T2D) is insufficient. The study group hypothesizes that a lower carbohydrate content in the diabetic diet than the recommended 55 energy percentage (E%) will decrease the postprandial glucose excursion. This will reduce postprandial insulin concentration, which together with lower glucose concentration leads to less fat accumulation in the liver and muscle tissue, resulting in an improved insulin sensitivity which together with a reduced glucose load improves the glucose metabolism. This clinical study will examine in subjects with type 2 diabetes the effect of highly controlled dietary low carbohydrate intervention on metabolic pathways with respect to insulin action, pancreatic islet function, lipid metabolism, ectopic fat accumulation, incretin hormones, low grade inflammation in plasma and adipose tissue, novel measures of fatty acid metabolism, and heart rate variability, respectively. The studies exhibit the potential to reform dietary recommendation aiming to prevent and ameliorate type 2 diabetes.

DETAILED DESCRIPTION:
The study will be performed as a randomized 12 weeks controlled, cross-over trial, which will address the effects on T2D of an isoenergetic low carbohydrate diet (carbohydrate 30 E%, protein 30 E%, fat 40 E%) compared to an isoenergetic control diet (carbohydrate 50 E%, protein 17 E%, fat 33 E%) currently recommended to individuals with T2D. The study is extended with 24 weeks on an isoenergetic low carbohydrate diet to examine the prolonged effect of the experimental diet on T2D and its pathophysiology. To test the hypothesis that the isoenergetic control diet is detrimental to glucose metabolism after only a short transition to this diet, the participants are reinforced to eat that diet during 6 weeks after the 24 weeks on low carbohydrate/high protein diet.

The study includes n=30 subjects with T2D. All study participants will be provided all meals for both the low carbohydrate diet and the control diet for free in the first part of the study, i.e. week 0 to 12, and these food items will be prepared and distributed from the research kitchen of the Department of Nutrition, Exercise and Sports, Faculty of Science, University of Copenhagen, Denmark to optimize compliance and adherence to the prescriped diet. During the isoenergetic diet study weight stability is reinforced to facilitate interpretation of the diet effect. All diets will be isoenergetic in accordance with the participant's estimated daily total energy expenditure (TEE). A dual energy X-ray absorptiometry (DXA) scan will be undertaken to determine body composition for each participant in order to estimate daily resting energy expenditure (REE). To estimate TEE, physical activity level expressed as PAL = TEE / REE, will be estimated. If a participant develops weight loss or weight gain at three consecutive measurements and/or lose or gain > 1kg of weight compared to baseline, the amount of energy in the diet wil be adjusted accordingly to enforce weight stability throughout the full duration of the study.

Measurements includes glycated hemoglobin (HbA1c) and fasting glucose, insulin, C-peptide and non-esterified fatty acids (NEFA) every 2 weeks during the first 12 weeks of the study and every 4 weeks from week 12.

At baseline, week 6, 12, 36 and 42, respectively larger measurement programs will be undertaken including insulin modified frequently sampled intravenous glucose tests (IM-FSIGT) and meal tests by use of Minimal Modelling, magnetic resonance imaging (MRi) for fat content in liver, abdomen and muscle, adipose tissue biopsies, continous glucose monitoring for 48-hours including diurnal blood pressure and Holter recording.

A standard meal will be provided for dinner a day prior to the measurement programs at week 0, 36 and 42. At weeks 6 and 12 the participants will intake their assigned meals. Participants will be informed to refrain from any strenuous physical activity and alcohol intake two days prior to and during the measurement program days.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed before any study-specific procedure
* Type 2 diabetes with glycated hemoglobin (HbA1c) between 48 mmol/mol and 97 mmol/mol with or without oral antidiabetic medicine
* Age > 18 years, men and women
* Hemoglobin > 7 mmol/L for men and > 6 mmol/L for women
* Estimated glomerular filtration rate (eGFR) > 30 mL/min/1.73 m2

Exclusion Criteria:

* Critical illness
* Systemic corticosteriod treatment e.g. prednisolone
* Reported or journalized severe food allergy or intolerance
* Reported or journalized severe gut disease e.g. Crohn's disease, Coeliac disease etc.
* Reported or journalized alcohol dependence syndrome
* Injectable diabetes medication
* Repeated fasting plasma glucose > 13.3 mmol/l
* Urine albumin / creatinine ratio > 300 mg/g
* Lactation, Pregnancy or planning of pregnancy during the study
* Inability, physically or mentally, to comply with the procedures required by the study protocol, as evaluated by the principal investigator
* Blood donation < 1 month prior to the study and during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-04; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Changes in glycated hemoglobin (HbA1c) at the end of 6 weeks of isoenergetic low carbohydrate diet compared to 6 weeks of the recommended antidiabetic control diet. | 42 weeks
  Changes in HbA1c during a fully controlled dietary cross-over intervention from baseline to week 6 will be compared to changes in HbA1c from week 6 to week 12. Changes in HbA1c will be assessed from week 12 to week 36 during a prolonged period where the participants receive dietician guidance to reinforce coherence to the low carbohydrate diet. HbA1c will be assessed at a follow-up visit at week 42. In addition HbA1c will be meassured every 14 days during the first 12 weeks, and every 4 weeks during the 24 weeks prolonged period. HbA1c will be expressed in mmol/mol.

SECONDARY OUTCOMES:
Changes in heart rate variability (HRV) from baseline to week 6 will be compared to changes in HRV from week 6 to 12. Changes in HRV will be assessed from week 12 to 36. | 36 weeks
  HRV will be assessed by a Holter monitor (model RZ 153+12 from Rozinn) at baseline, week 6, 12 and 36.
Changes in diurnal blood pressure (DBP) from baseline to week 6 will be compared to changes in DBP from week 6 to 12. Changes in DBP will be assessed from week 12 to 36. | 36 weeks
  DBP will be assessed by a blood pressure monitor (model 90217 from Spacelabs Healthcare) at baseline, week 6, 12 and 36.
Changes in insulin sensitivity from baseline to week 6 will be compared to changes in insulin sensitivity from week 6 to 12. Changes in insulin sensitivity will be assessed from week 12 to 36. | 36 weeks
  Changes in insulin sensitivity will be measured using the minimal model technique based on a insulin modified frequently sample intravenous glucose test (IM-FSIGT) at baseline, week 6, 12 and 36.
Changes in beta-cell function from baseline to week 6 will be compared to changes in beta-cell function from week 6 to 12. Changes in beta-cell function will be assessed from week 12 to 36. | 36 weeks
  Changes in beta-cell function will be measured using the minimal model technique based on a insulin modified frequently sample intravenous glucose test (IM-FSIGT) at baseline, week 6, 12 and 36.
Changes in glucagon-like-petide-1 (GLP-1) at baseline to week 6 will be compared to changes in GLP-1 from week 6 to 12. Changes in GLP-1 will be assessed from week 12 to 36. | 36 weeks
  Changes in GLP-1 will be measured during a 4-hour (4-h) mixed meal test (MMT) at baseline, week 6, 12 and 36. GLP-1 will be expressed in pmol/L.
Changes in glucose-dependent insulinotropic polypeptide (GIP) at baseline to week 6 will be compared to changes in GIP from week 6 to 12. Changes in GIP will be assessed from week 12 to 36. | 36 weeks
  Changes in GIP will be measured during a 4-h MMT at baseline, week 6, 12 and 36. GIP will be expressed in pmol/L.
Changes in insulin-like growth factor-1 (IGF-1) at baseline to week 6 will be compared to changes in IGF-1 from week 6 to 12. Changes in IGF-1 will be assessed from week 12 to 36. | 36 weeks
  Changes in IGF-1 will be measured during a 4-h MMT at baseline, week 6, 12 and 36. IGF-1 will be expressed in ng/mL.
Changes in insulin-like growth factor-binding protein 1 (IGFBP-1) at baseline to week 6 will be compared to changes from week 6 to 12. Changes in IGFBP-1 will be assessed from week 12 to 36. | 36 weeks.
  Changes in IGFBP-1 will be measured during a 4-h MMT at baseline, week 6, 12 and 36. IGFBP-1 will be expressed in ng/mL.
Changes in growth hormone (GH) at baseline to week 6 will be compared to changes in GH from week 6 to 12. Changes in GH will be assessed from week 12 to 36. | 36 weeks.
  Changes in GH will be measured during a 4-h MMT at baseline, week 6, 12 and 36. GH will be expressed in ng/mL.
Changes in colecystokinin (CCK) at baseline to week 6 will be compared to changes in CCK from week 6 to 12. Changes in CCK will be assessed from week 12 to 36. | 36 weeks
  Changes in CCK will be measured during a 4-h MMT at baseline, week 6, 12 and 36. CCK will be expressed as pmol/L.
Changes in peptide YY (PYY) at baseline to week 6 will be compared to changes in PYY from week 6 to 12. Changes in PYY will be assessed from week 12 to 36. | 36 weeks
  Changes in PYY will be measured during a 4-h MMT at baseline, week 6, 12 and 36. PYY will be expressed as pmol/L.
Changes in ghrelin at baseline to week 6 will be compared to changes in ghrelin from week 6 to 12. Changes in ghrelin will be assessed from week 12 to 36. | 36 weeks
  Changes in ghrelin will be measured during a 4-h MMT at baseline, week 6, 12 and 36. Ghrelin will be expressed as pmol/L.
Changes in liver, skeletal muscle and visceral fat composition will be compared to changes in fat composition from week 6 to 12. Changes in fat composition will be assessed from week 12 to 36. | 36 weeks
  Changes in liver, skeletal muscle and visceral adipose tissue will be assessed by magnetic resonance imaging (MRi) at baseline, week 6, 12 and 36.
Changes in subjective satiety at baseline to week 6 will be compared to changes subjective satiety from week 6 to 12. Changes in subjective satiety will be assessed from week 12 to 36. | 36 weeks.
  Changes in subjective satiety will be assessed by a self-reported visual analog scale (VAS) questionnaire in relation to a 4-h MMT at baseline, week 6, 12 and 36.
Changes in anxiety and depression symptoms at baseline to week 6 compared to changes from week 6 to 12. Changes in anxiety and depression symptoms will be assessed at week 12 to 36. | 36 weeks.
  Changes will be assessed by a self-reported hospital anxiety and depression scale (HADS) questionnaire at baseline, week 6, 12 and 36.
Changes in insulin at baseline to week 6 will be compared to changes in insulin from week 6 to 12. Changes in insulin will be assessed from week 12 to 36. | 36 weeks.
  Changes in insulin will be assessed during a 4-h MMT and during a IM-FSIGT-test at baseline, week 6, 12 and 36. In addition insulin will be meassured every 14 days during the first 12 weeks, and every 4 weeks during the last 24 weeks. Insulin will be expressed in pmol/L.
Changes in C-peptide at baseline to week 6 will be compared to changes in C-peptide from week 6 to 12. Changes in C-peptide will be assessed from week 12 to 36. | 36 weeks.
  Changes in C-peptide will be assessed during a 4-h MMT and during a IM-FSIGT-test at baseline, week 6, 12 and 36. In addition C-peptide will be measured every 14 days during the first 12 weeks, and every 4 weeks during the last 24 weeks. C-peptide will be expressed in pmol/L.
Changes in non-esterified fatty acids (NEFA) at baseline to week 6 will be compared to changes in NEFA from week 6 to 12. Changes in NEFA will be assessed from week 12 to 36. | 36 weeks.
  Changes in NEFA will be assessed during a 4-h MMT and during a IM-FSIGT-test at baseline, week 6, 12 and 36. In addition NEFA will be meassured every 14 days during the first 12 weeks, and every 4 weeks during the last 24 weeks. NEFA will be expressed in micromol/L.
Changes in blood glucose at baseline to week 6 will be compared to changes in blood glucose from week 6 to 12. Changes in blood glucose will be assessed from week 12 to 36. | 36 weeks
  Changes in blood glucose will be assessed during a 4-h MMT and during a IM-FSIGT-test at baseline, week 6, 12 and 36. Blood glucose will be expressed as mmol/L.
Changes in insulin-like growth factor-binding protein 3 (IGFBP-3) at baseline to week 6 will be compared to changes from week 6 to 12. Changes in IGFBP-3 will be assessed from week 12 to 36. | 36 weeks.
  Changes in IGFBP-1 will be measured during a 4-h MMT at baseline, week 6, 12 and 36. IGFBP-1 will be expressed in ng/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Thure Krarup, MD, DMSc, Study Director — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomsen MN, Skytte MJ, Samkani A, Weber P, Fenger M, Frystyk J, Hansen E, Holst JJ, Madsbad S, Magkos F, Thomsen HS, Walzem RL, Haugaard SB, Krarup T. Replacing dietary carbohydrate with protein and fat improves lipoprotein subclass profile and liver fat in type 2 diabetes independent of body weight: evidence from 2 randomized controlled trials. Am J Clin Nutr. 2025 Feb;121(2):224-231. doi: 10.1016/j.ajcnut.2024.11.030. Epub 2024 Nov 29. PMID 39617302
- [Derived] Alzahrani AH, Skytte MJ, Samkani A, Thomsen MN, Astrup A, Ritz C, Chabanova E, Frystyk J, Holst JJ, Thomsen HS, Madsbad S, Haugaard SB, Krarup T, Larsen TM, Magkos F. Body weight and metabolic risk factors in patients with type 2 diabetes on a self-selected high-protein low-carbohydrate diet. Eur J Nutr. 2021 Dec;60(8):4473-4482. doi: 10.1007/s00394-021-02605-0. Epub 2021 Jun 8. PMID 34101004
- [Derived] Skytte MJ, Samkani A, Petersen AD, Thomsen MN, Astrup A, Chabanova E, Frystyk J, Holst JJ, Thomsen HS, Madsbad S, Larsen TM, Haugaard SB, Krarup T. A carbohydrate-reduced high-protein diet improves HbA1c and liver fat content in weight stable participants with type 2 diabetes: a randomised controlled trial. Diabetologia. 2019 Nov;62(11):2066-2078. doi: 10.1007/s00125-019-4956-4. Epub 2019 Jul 23. PMID 31338545